CLINICAL TRIAL: NCT02976025
Title: Remote Supervision for Implementing Collaborative Care for Perinatal Depression
Acronym: MInD-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: OCHIN, Inc. (Other); Oregon Social Learning Center (Other); University of Pennsylvania (Other); Washington University School of Medicine (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ian Bennett, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001294; 1R01MH108548-01 (NIH)
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Perinatal Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Longitudinal Remote Consultation (Experimental): This is the active treatment arm consisting of 10 cluster randomized health centers receiving both training in collaborative care and longitudinal remote consultation (LRC) support.
  Interventions: Other: Longitudinal Remote Consultation
- Collaborative Care (Active Comparator): This comparator arm will consist of 10 cluster randomized health centers who receive training in collaborative care.
  Interventions: Other: Collaborative Care

INTERVENTIONS:
Other: Longitudinal Remote Consultation — Longitudinal Remote Consultation utilizes video conferencing to efficiently link providers to consultants who provide timely feedback and training in collaborative care. LRC will be provided in addition to standard collaborative care training and support.
  Other Names: LRC
  Arms: Longitudinal Remote Consultation
Other: Collaborative Care — Standard collaborative care implementation training and support.
  Other Names: CC
  Arms: Collaborative Care

SUMMARY:
This study evaluates the impact of a longitudinal remote consultation (LRC) implementation strategy for collaborative care depression treatment among perinatal women. All participating health centers will receive training in collaborative care. Cluster randomization will be used to assign the addition of LRC to select health centers. Differences in implementation success, clinical outcomes, and costs will be compared after a 12 month implementation period and 13-21 month sustainment period.

DETAILED DESCRIPTION:
Depression is a common and serious disorder among pregnant women but few from low income groups receive effective treatment. The highly evidence based collaborative care (CC) model for depression has been shown to work for women in pregnancy but has not been widely implemented in this population. The proposed study targets improving dissemination of the evidence based CC treatment model for pregnant and postpartum women with depression, a common disorder of the perinatal period (pregnancy and the first year following birth). Longitudinal remote consultation (LRC) is an implementation strategy that has been have shown to improve fidelity to evidence-based practices and patient outcomes for mental health innovations. The investigators believe LRC can be used with equal benefit for complex interventions such as CC.

The purpose of this study is to compare two implementation strategies for Collaborative Care depression treatment: 1) standard implementation and 2) standard implementation + Longitudinal Remote Consultation (LRC). This research is being done in order to assess implementation and patient outcomes in sites receiving a standard implementation approach with and without LRC. The results of the proposed study will provide information on the benefits and relative value of ongoing consultation, such as LRC, for implementation of complex interventions like collaborative care.

The proposed study will involve twenty health centers providing prenatal care which are part of the national OCHIN Network or other health center network. All sites will receive a standard implementation approach. After pre-implementation training ten of the sites will be randomly selected to receive LRC. Implementation and clinical outcomes as well as costs will be compared between the study conditions after a 12 month implementation period and a 13-21 month sustainment period. The results of the proposed study will provide critical generalizable knowledge regarding the benefits of ongoing consultation for implementation of complex interventions like collaborative care.

ELIGIBILITY:
Patient Participants:

Inclusion Criteria:

* Patient participants must be perinatal women,
* Age 18-45,
* Receiving care at one of the 20 OCHIN or non-OCHIN health centers participating in the study and must have major depression as determined by a score of ≥10 on the PHQ-9 depression screener.

Exclusion Criteria:

* Age <18 or >45,
* Male.

Health Center Participating Sites:

Inclusion Criteria:

* Use of the shared OCHIN Epic electronic record for perinatal care or use of the secure AIMS CMTS/Caseload Tracker/spreadsheet patient registry for perinatal care and
* A minimum of 50 prenatal patients annually.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Clinical depression outcomes | 12 months post-initiation of collaborative care
  Patient Health Questionnaire-9 (PHQ-9); level of depression symptomatology and functional impairment.

SECONDARY OUTCOMES:
Implementation outcomes | 12 month post-implementation of collaborative care
  To assess the degree to which sites in the two conditions complete implementation, the investigators will use the Stages of Implementation Completion tool tailored for collaborative care, SIC-CC.

OTHER OUTCOMES:
Cost and cost-effectiveness | 12-month post-implementation of collaborative care
  For a cost-benefit analysis, the investigators will use of the Cost of Implementing New Strategies (COINS) method to assess costs in the two conditions. This methodology takes advantage of the SIC-CC instrument as a costing template to map the use of resources and associated costs to these to study conditions. Costs associated with implementation in each of these conditions will be carried out for all 20 health centers included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Bennett, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We intend to share de-identified data once study is complete.

REFERENCES:
- [Derived] Grover T, Bennett IM, Campbell M, Vredevoogd M, Saldana L. Implementation cost analysis of collaborative care for perinatal mental health in community health centers. Res Sq [Preprint]. 2024 Nov 27:rs.3.rs-5256122. doi: 10.21203/rs.3.rs-5256122/v1. PMID 39649162